CLINICAL TRIAL: NCT02464800
Title: Efficacy of Higher Cutting Rate in Microincision Vitrectomy for Proliferative Diabetic Retinopathy
Status: Completed | Type: Observational
Sponsor: Kyorin University (Other)
Responsible Party: Principal Investigator, Makoto Inoue, Kyorin Eye center, Kyorin University
Other Study IDs: Kyorineye016
Record Dates: First submitted 2015-06-02; First posted 2015-06-08 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Proliferative Diabetic Retinopathy
Keywords: diabetic retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Vitrectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Higher cutting rate group: Vitrectomy with higher cutting rate instruments (5000 cut per minute) were performed in 174 eyes for proliferative diabetic retinopathy
  Interventions: Procedure: Vitrectomy for proliferative diabetic retinopathy
- Conventional cutting rate group: Vitrectomy with conventional instruments (2500 cut per minute) were performed in 219 eyes for proliferative diabetic retinopathy
  Interventions: Procedure: Vitrectomy for proliferative diabetic retinopathy

INTERVENTIONS:
Procedure: Vitrectomy for proliferative diabetic retinopathy — 25-gauge vitrectomy

SUMMARY:
The medical records of 393 eyes of 326 patients with severe proliferative diabetic retinopathy were reviewed. Higher cutting rate instruments (5000 cut per minute) were used in 174 eyes and conventional instruments in 219 eyes (2500 cut per minute). The visual outcome and incidences of intraoperative and postoperative complications were compared.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were patients who had persistent vitreous hemorrhage, fibrovascular proliferation affecting the macula, or tractional RD and who had a follow-up for more than 6 months.

Exclusion Criteria:

* The eyes with follow-up less than 6 months

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who underwent 25-gauge vitrectomy for proliferative diabetic retinopathy with higher cutting rate instruments or conventional instruments
Sampling Method: Non-Probability Sample
Enrollment: 326 (Actual)
Dates: Start 2007-04; Primary Completion 2014-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 6 months

SECONDARY OUTCOMES:
Retinal reattachment | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Makoto Inoue, Mitaka, Tokyo, Japan